CLINICAL TRIAL: NCT03052283
Title: Evaluation and Validation of a New Questionnaire to Identify and Quantify Abdominal Symptoms in Patients With Cystic Fibrosis Following FDA Guidelines: the CF Abd-Score (Primarily Named JenAbdomen-CF Score)
Brief Title: Development and Validation of a Disease Specific PROM to Assess Abdominal Involvement in Patients With CF (CFAbd-Score)
Acronym: CFAbd-Score
Status: Recruiting | Type: Observational
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Collaborators: University of Jena (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jochen G. Mainz, Director of the Cystic Fibrosis-Center, Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: CFAbd-Score; CFAbd-Score.kid (Other: Brandenburg Med.School (Univ.), Brandenb.a.d.Havel/Germany); CFAbd-day2day (Other: Brandenburg Med.School (Univ.), Brandenb.a.d.Havel/Germany)
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Abdomen; Pancreas; Liver; Gut; Symptom Score; Patient reported outcome measure (PROM); diabetes; CFTR-modulator; Tricafta; Kaftrio
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CF: >2000 in Germany, France, Italy, Spain, Denmark, Belgium, Portugal, GB, Ireland, USA, Australia, Canada, Brazil, Argentina...
  Interventions: Diagnostic Test: Questionnaire Patient Reported Outcome Measure (PROM)
- Age-matched healthy controls: >100 in Germany >100 in each of the other participating countries
  Interventions: Diagnostic Test: Questionnaire Patient Reported Outcome Measure (PROM)

INTERVENTIONS:
Diagnostic Test: Questionnaire Patient Reported Outcome Measure (PROM) — non-interventional
  Other Names: routine-care assessments

SUMMARY:
Development, validation and evaluation of a new multimodal questionnaire to assess and quantify the abdominal involvement in patients with the inherited life shortening multi-organ disease Cystic fibrosis.

In the stepwhise development of the patient reported outcome measures (PROM) repeadedly, CF-patients, their families as well as professionals working in different fields of CF-care will be included.

DETAILED DESCRIPTION:
Development of a multimodal questionnaire considering the FDA guidelines for development of a PROM, the CFAbd-Score

* Evaluation of reliability of the questionnaire by examining internal consistency and construct validity
* Evaluation of reproducibility of the questionnaire by re-testing of patients
* Assessment of cross-generational applicability of the questionnaire by sub-scoring of age groups
* Evaluation of the responsiveness of the score by comparison with age-matched healthy controls
* Assessment of putative relationships of abdominal symptoms with faecal inflammatory markers
* Assessment of applicability of the questionnaire in other CF centers
* Transfer the CFAbd-Score to other countries and languages

Development and validation of a CF-specific tool for daily assessment of abdominal symptoms (patient diary), the CFAbd-day2day

Development and validation of a CF-specific tool for assessment of abdominal symptoms in children < 12 years of age, the CFAbd-kid

ELIGIBILITY:
Inclusion Criteria:

CF cohort:

Diagnosis of CF determined by

* a sweat chloride of >60 mEq/L and/or
* detection of 2 disease causing CFTR mutations with evidence of organ involvement.

Healthy controls:

* Age-matched

Exclusion Criteria:

CF cohort:

* Lacking ability to cooperate of patients /their families, respectively

Healthy controls:

* Other diseases causing abdominal symptoms (Inflammatory bowel disease (IBD), alpha 1 antitrypsin deficiency, celiac disease, food allergy, gastroenteritis, etc.)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CF of all ages
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-01-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Development and evaluation of the CFAbd-Score (initially named JenAbdomen CF-Score), a CF-specific PROM following FDA recommendations | 7 years
  Evaluation and validation of the CFAbd-Score based on a CF patient-reported outcome measure (PROM) that includes all relevant gastrointestinal symptoms and their impact on subjective quality of life
Development and evaluation of a diary for assessment and quantification of abdominal symptoms, a CF-specific PROM following FDA recommendations | 7

SECONDARY OUTCOMES:
Abdominal symptoms in cystic fibrosis and their relation to genotype, history, clinical and laboratory findings | 7 years
  relating CFAbd-Scores to history, clinical- and laboratory findings
Assessing the Relation of Ultrasound Findings and Abdominal Symptoms obtained with the CFAbd-Score in Cystic Fibrosis Patients | 3 years
  abdominal ultrasound
Effects of a new therapy with CFTR-modulator on abdominal symtoms, quantified with the CFAbd-Score | 7 years
  Assessing the CFAbd-Score´s sensitivity to identify and quantify changes due to effective therapeutic interventions, following FDA-guidelines for validation of a PROM

CONTACTS AND LOCATIONS:
Overall Officials: Jochen G Mainz, Prof. MD, Principal Investigator — Medizinische Hochschule Brandenburg (MHB), University
Locations (2):
- Germany (2):
  - Klinikum Westbrandenburg, Brandenburg
  - Medizinische Hochschule Brandenburg (MHB), University, Brandenburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tabori H, Arnold C, Jaudszus A, Mentzel HJ, Renz DM, Reinsch S, Lorenz M, Michl R, Gerber A, Lehmann T, Mainz JG. Abdominal symptoms in cystic fibrosis and their relation to genotype, history, clinical and laboratory findings. PLoS One. 2017 May 4;12(5):e0174463. doi: 10.1371/journal.pone.0174463. eCollection 2017. PMID 28472055
- [Result] Tabori H, Jaudszus A, Arnold C, Mentzel HJ, Lorenz M, Michl RK, Lehmann T, Renz DM, Mainz JG. Relation of Ultrasound Findings and Abdominal Symptoms obtained with the CFAbd-Score in Cystic Fibrosis Patients. Sci Rep. 2017 Dec 12;7(1):17465. doi: 10.1038/s41598-017-17302-4. PMID 29234058
- [Result] Jaudszus A, Zeman E, Jans T, Pfeifer E, Tabori H, Arnold C, Michl RK, Lorenz M, Beiersdorf N, Mainz JG. Validity and Reliability of a Novel Multimodal Questionnaire for the Assessment of Abdominal Symptoms in People with Cystic Fibrosis (CFAbd-Score). Patient. 2019 Aug;12(4):419-428. doi: 10.1007/s40271-019-00361-2. PMID 30887269
- [Result] Jaudszus A, Pfeifer E, Lorenz M, Beiersdorf N, Hipler UC, Zagoya C, Mainz JG. Abdominal Symptoms Assessed With the CFAbd-Score are Associated With Intestinal Inflammation in Patients With Cystic Fibrosis. J Pediatr Gastroenterol Nutr. 2022 Mar 1;74(3):355-360. doi: 10.1097/MPG.0000000000003357. PMID 34789668
- [Result] Mainz JG, Zagoya C, Polte L, Naehrlich L, Sasse L, Eickmeier O, Smaczny C, Barucha A, Bechinger L, Duckstein F, Kurzidim L, Eschenhagen P, Caley L, Peckham D, Schwarz C. Elexacaftor-Tezacaftor-Ivacaftor Treatment Reduces Abdominal Symptoms in Cystic Fibrosis-Early results Obtained With the CF-Specific CFAbd-Score. Front Pharmacol. 2022 Jun 3;13:877118. doi: 10.3389/fphar.2022.877118. eCollection 2022. PMID 35721187
- [Result] Caley LR, Zagoya C, Duckstein F, White H, Shimmin D, Jones AM, Barrett J, Whitehouse JL, Floto RA, Mainz JG, Peckham DG. Diabetes is associated with increased burden of gastrointestinal symptoms in adults with cystic fibrosis. J Cyst Fibros. 2023 Mar;22(2):275-281. doi: 10.1016/j.jcf.2023.01.010. Epub 2023 Jan 27. PMID 36710099
- See also: Validity and Reliability of a Novel Multimodal Questionnaire for the Assessment of Abdominal Symptoms in People with Cystic Fibrosis (CFAbd-Score). — https://link.springer.com/article/10.1007%2Fs40271-019-00361-2